CLINICAL TRIAL: NCT04390308
Title: Is There A Role For Mechanical Stimulation In Ovarian Follicular Activation? A Randomized Control Trial.
Brief Title: Is There A Role For Mechanical Stimulation In Ovarian Follicular Activation?
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2004-ABU-005-LM
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female; Premature Ovarian Failure; IVF
MeSH Terms: conditions — Infertility, Female; Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: The cortex of selected ovary will be punctured up to ten times. In the surgical report, the surgeon will state how many punctures have been done.
  Interventions: Procedure: Ovarian puncture; Other: Hormonal blood Test; Diagnostic Test: Transvaginal ultrasound
- Control: No intervention

INTERVENTIONS:
Procedure: Ovarian puncture — Egg collection
  Groups: Intervention
Other: Hormonal blood Test — AMH (ng/ml), FSH (IU/mL), E2(pg/mL), P4(ng/mL), LH (IU/mL)
  Groups: Intervention
Diagnostic Test: Transvaginal ultrasound — Doppler of arteria ovarica. Resistance index
  Groups: Intervention

SUMMARY:
Premature ovarian failure (POI) is a loss of normal function before age 40, leading to infertility and hypoestrogenism. About 1% of women younger than 40 years old and 0.1% before 30 are affected. Most patients already had impaired or complete loss of fecundity when diagnosed. Hence, the treatment of POI is particularly tough. Currently, no optimal regimen exists to ameliorate ovarian function.

DETAILED DESCRIPTION:
In women, the non-growing population of follicles that comprise the ovarian reserve is determined at birth and serves as the reservoir for future fertility. This reserve of dormant, primordial follicles and the mechanisms controlling their selective activation which constitute the committing step into folliculogenesis are essential for determining fertility outcomes in women.

While POI is sometimes called premature menopause, it is not identical with menopause. Women with POI may still have occasional irregular periods and may even occasionally achieve a pregnancy. Symptoms of POI include irregular menses or amenorrhea, infertility, hypoestrogenic symptoms and decreased libido. POI may be caused by chromosomal defects such as mosaic Turner's syndrome, exposure to toxins (chemotherapy or radiation), autoimmunity, genetic factors (FMR1) and other unknown factors.

Recently, new promising approaches have emerged for infertility treatment in patients with POI, which are based on arousing the still available primordial follicle pool. It is supposed that these techniques activate dormant primordial follicles using a combination of mechanical signaling and biochemical factors. The hypothesis that mild local ovarian injury, such as ovarian puncture, which is a usual procedure in an IVF center with minimal side effects, might exert a similar favorable effect in women with POI arouses our curiosity.

Different groups have published case series of ovarian procedures, injecting substances in the ovaries (A-PRP) or ovarian biopsies / scratch in infertile patients with low ovarian reserve (LOR) or/and patients with POF. However, those studies were underpowered, including not enough number of cases, with variable inclusion criteria and reporting results with very low scientific evidence. Furthermore, the mechanical effect of injecting the ovary should be taken into consideration during the evaluation of these patients, yet it might improve the ovarian function as well.

There are no previous randomized controlled trials considering a procedure as ovarian puncture, which is easier and accessible at any fertility center.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women 40 years of age and younger with documented primary ovarian insufficiency (12).
* Normal Karyotype
* BMI </= 35 kg/m2
* Oligo/amenorrhea for at least 4 months
* FSH > 25 IU/mL
* AMH </= 0,1 ng/ml
* No evidence of follicles > 4mm
* Must have two ovaries of approximately equal volume.
* Willingness to undergo further fertility treatment, including IVF if there is evidence of response
* A transvaginal scan including Doppler for arteria ovarica will be performed previously to the surgical procedure.

Exclusion Criteria:

* Premature ovarian failure due to a genetic origin, such as Turner's Syndrome or chromosomal abnormality.
* Oncological diseases (specially, skeletal system and blood).
* Autoimmune diseases, for example, lupus erythematosus, etc.
* Previous treatments including radiotherapy or chemotherapy.
* Other conditions not suitable for surgical procedures and/or anesthesia.
* Anticoagulant or antiaggregant treatment.
* Acute and chronic infectious diseases.
* Active substance abuse or dependence.
* Major Mental health disorder.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Adult women with primary or secondary infertility with a diagnosis of POI, willing to perform an IVF treatment
Study Population: Adult women with primary or secondary infertility with a diagnosis of POI, willing to perform an IVF treatment
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Follicle growth above 4 mm | 1 day
  One or more follicles evaluated by transvaginal ultrasound. Defined by number of follicles growing, quantitative variable.
Anti-Müllerian hormone evaluation after intervention. | 1 day
  Anti-Müllerian hormone evaluation after intervention.
Follicle-stimulating hormone evaluation after intervention. | 1 day
  Follicle-stimulating hormone evaluation after intervention.
Luteinizing hormone evaluation after intervention. | 1 day
  Luteinizing hormone evaluation after intervention.
Estradiol hormone evaluation after intervention. | 1 day
  Estradiol hormone evaluation after intervention.
Progesterone hormone evaluation after intervention. | 1 day
  Progesterone hormone evaluation after intervention.
Spontaneous menstruation. | 1 day
  Spontaneous menstruation.
Arteria ovarica doppler results. | 1 day
  Arteria ovarica doppler results. Resistance index.

SECONDARY OUTCOMES:
Number of follicles | 1 day
  Number of follicles
Number of oocytes retrieved | 1 day
  Number of oocytes retrieved
Fertilization rate | 1 day
  percentage of 2PN embryos per oocyte injected
Blastulation rate | 1 day
  percentage of blastocysts per 2PN embryos
Aneuploidy rate | 1 day
  percentage of aneuploid blastocysts per total blastocyst biopsied

OTHER OUTCOMES:
Clinical pregnancy by blood test | 12 weeks
  pregnancy (yes or no) defined by a βhCG test of > 15IU
Implantation rate (%) | 4 weeks
  defined by the number of gestational sacs/number of embryos transferred
Clinical pregnancy by ultrasound | 12 weeks
  defined by the ultrasonographic visualization of one or more gestational sacs, including ectopic pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Laura Melado, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ford EA, Beckett EL, Roman SD, McLaughlin EA, Sutherland JM. Advances in human primordial follicle activation and premature ovarian insufficiency. Reproduction. 2020 Jan;159(1):R15-R29. doi: 10.1530/REP-19-0201. PMID 31376814
- [Background] Zhang X, Han T, Yan L, Jiao X, Qin Y, Chen ZJ. Resumption of Ovarian Function After Ovarian Biopsy/Scratch in Patients With Premature Ovarian Insufficiency. Reprod Sci. 2019 Feb;26(2):207-213. doi: 10.1177/1933719118818906. Epub 2018 Dec 12. PMID 30541396
- [Background] Kawamura K, Kawamura N, Hsueh AJ. Activation of dormant follicles: a new treatment for premature ovarian failure? Curr Opin Obstet Gynecol. 2016 Jun;28(3):217-22. doi: 10.1097/GCO.0000000000000268. PMID 27022685
- [Background] Nurden AT. Platelets, inflammation and tissue regeneration. Thromb Haemost. 2011 May;105 Suppl 1:S13-33. doi: 10.1160/THS10-11-0720. Epub 2011 Apr 11. PMID 21479340
- [Background] Gurtner GC, Werner S, Barrandon Y, Longaker MT. Wound repair and regeneration. Nature. 2008 May 15;453(7193):314-21. doi: 10.1038/nature07039. PMID 18480812
- [Background] Lacci KM, Dardik A. Platelet-rich plasma: support for its use in wound healing. Yale J Biol Med. 2010 Mar;83(1):1-9. PMID 20351977
- [Background] Sfakianoudis K, Simopoulou M, Nitsos N, Rapani A, Pantou A, Vaxevanoglou T, Kokkali G, Koutsilieris M, Pantos K. A Case Series on Platelet-Rich Plasma Revolutionary Management of Poor Responder Patients. Gynecol Obstet Invest. 2019;84(1):99-106. doi: 10.1159/000491697. Epub 2018 Aug 22. PMID 30134239
- [Background] Sills ES, Rickers NS, Li X, Palermo GD. First data on in vitro fertilization and blastocyst formation after intraovarian injection of calcium gluconate-activated autologous platelet rich plasma. Gynecol Endocrinol. 2018 Sep;34(9):756-760. doi: 10.1080/09513590.2018.1445219. Epub 2018 Feb 28. PMID 29486615
- [Background] Sills ES, Li X, Rickers NS, Wood SH, Palermo GD. Metabolic and neurobehavioral response following intraovarian administration of autologous activated platelet rich plasma: First qualitative data. Neuro Endocrinol Lett. 2019 Jan;39(6):427-433. PMID 30796792
- [Background] Sills ES, Rickers NS, Svid CS, Rickers JM, Wood SH. Normalized Ploidy Following 20 Consecutive Blastocysts with Chromosomal Error: Healthy 46, XY Pregnancy with IVF after Intraovarian Injection of Autologous Enriched Platelet-derived Growth Factors. Int J Mol Cell Med. 2019 Winter;8(1):84-90. doi: 10.22088/IJMCM.BUMS.8.1.84. Epub 2019 May 15. PMID 32195207
- [Background] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- See also: Ovarian rejuvenation and folliculogenesis reactivation in peri-menopausal women after autologous platelet-rich plasma treatment — https://sa1s3.patientpop.com/assets/docs/111052.pdf